CLINICAL TRIAL: NCT07183748
Title: A Double-blind, Phase II Feasibility Study to Assess the Safety and Efficacy of Psilocybin Microdosing Combined With Psychotherapy in Treatment-resistant Depression
Brief Title: Psilocybin Microdosing With Psychotherapy for Treatment-Resistant Depression
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beersheva Mental Health Center (Other Government)
Collaborators: MSICS PHARMA LTD (Unknown)
Responsible Party: Principal Investigator, ODED ARBEL, Principal Investigator, Beersheva Mental Health Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MHC-5-22
Record Dates: First submitted 2025-06-15; First posted 2025-09-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-08

CONDITIONS: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Psilocybin; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Drug: Psilocybin (drug)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Psilocybin (drug) — 0.4 grams
  Arms: Treatment
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Objective:

To assess the safety and efficacy of a six-week microdosing regimen of psilocybin combined with short-term, experience-based psychotherapy in patients with treatment-resistant depression who have not responded to previous pharmacological or long-term psychological interventions.

Hypothesis:

Compared to baseline, the group that begins with psilocybin will exhibit a more rapid reduction in depressive symptoms after six weeks, compared to the group that begins with placebo and receives only psychotherapy. Following the crossover between conditions, the placebo-first group will also show an accelerated reduction in these measures after the subsequent six weeks.

Alternative hypothesis: No difference will be observed between groups in the rate of symptom reduction.

Objective:

To examine biological markers that may mediate potential improvements in depressive symptoms among participants receiving psilocybin microdosing compared to placebo.

Hypothesis:

Compared to baseline, six weeks of active psilocybin dosing will result in decreased levels of cortisol and inflammatory markers, and increased levels of oxytocin and BDNF in saliva.

Objective:

To assess psychological factors that may mediate potential improvements in depressive symptoms among participants receiving psilocybin microdosing compared to placebo.

Hypothesis:

Compared to baseline, six weeks of active psilocybin dosing will lead to increased cognitive flexibility, greater self-compassion, and enhanced present-moment awareness.

Objective:

To explore a subpopulation of women experiencing premenstrual symptom exacerbation (PMS) and the potential for improvement in depressive symptoms in the days preceding menstruation, if any.

Hypothesis:

Among women with worsened premenstrual symptoms, psilocybin will reduce premenstrual symptoms, specifically depressive symptoms, compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 18-65 years.
* Diagnosis of treatment-resistant major depression as defined by the DSM-IV criteria (309.81) (ASA 1994) and determined by the BDI (BDI-II, 1996).
* Willingness to discontinue psychiatric medication starting two weeks prior to the beginning of the study and throughout its duration, as well as to cease the use of drugs and licensed cannabis, and to suspend psychotherapy for the duration of the study. Participants also commit not to initiate psychiatric medication or psychotherapy during the study without consulting the research team. All under supervision within a day treatment framework.
* Abstinence from drugs and other psychiatric medications.
* Negative pregnancy test for women, and use of contraception by both men and women during the study period.
* Willingness to sign a confidentiality waiver allowing the research team to consult with the participant's treating physician.
* Willingness to provide the contact information of a close and relevant person in case suicidal ideation arises.
* Commitment to participate in all stages of the study, including follow-up assessments.
* Willingness not to participate in another study during the current study period.

Exclusion Criteria:

* Investigators and their immediate family members are not permitted to participate in the study. Immediate family is defined as the investigator's spouse, parent, child, grandparent, or grandchild.
* Pregnant women, breastfeeding women, or women of childbearing age who are not using medically approved contraceptive methods (e.g., condoms).

Men who are sexually active and may cause pregnancy but are unwilling to use contraception.

* Significant unstable physical illness (including cardiac, hepatic, renal, respiratory, endocrinological, neurological, or hematological conditions), based on the investigator's judgment.
* Psychotic spectrum disorders.
* Bipolar disorder.
* Post-traumatic disorder involving dissociative symptoms.
* Uncontrolled anxiety disorder.
* Chronic perceptual disorder (HPPD).
* Head injury or cognitive impairment (including intellectual disability or dementia).
* Severe suicidal risk or aggressive behavior toward others, as assessed by the investigator and standardized depression/suicide assessment questionnaires.

History of chronic benzodiazepine use (at least 4 mg lorazepam daily for over two years), or signs and symptoms of benzodiazepine use within two weeks prior to randomization.

* Alcohol and/or substance abuse within the past 6 months, based on the clinical judgment of the investigator.
* Any active addiction (substance use disorder).
* Current or past epilepsy.
* Individuals with focal or generalized encephalopathy (e.g., tumor, stroke, meningitis, encephalitis), or head trauma that may be epileptogenic.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory -II (BDI-II) change from baseline | Baseline, Weeks 2, 4, 6, 8, 10, 12, and 24
  depression symptoms, will be measured by the Beck Depression Inventory
Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline, Weeks 2, 4, 6, 8, 10, 12, and 24
  A standardized questionnaire that assesses suicidal ideation and behavior, including severity and intensity of thoughts, and history of suicide attempts.
Mindful Attention Awareness Scale (MAAS | Baseline, Weeks 2, 4, 6, 8, 10, 12, and 24
  A self-report questionnaire that measures the frequency of mindful states in day-to-day life, focusing on present-moment awareness and attention.
Five Facet Mindfulness Questionnaire (FFMQ) | Baseline, Weeks 2, 4, 6, 8, 10, 12, and 24
  A self-report measure that assesses five aspects of mindfulness: observing, describing, acting with awareness, non-judging, and non-reactivity.
Self-Compassion Scale, Neff, 2003b | Baseline, Weeks 2, 4, 6, 8, 10, 12, and 24
  self-report questionnaire that measures levels of self-compassion across dimensions such as self-kindness, common humanity, and mindfulness.
The Quality of Life Enjoyment & Satisfaction Questionnaire (Q-LESQ-SF) . | Baseline, Weeks 2, 4, 6, 8, 10, 12, and 24
  A self-report measure that evaluates an individual's degree of enjoyment and satisfaction in various areas of daily functioning and overall quality of life.
Premenstrual symptoms screening tool: PSST, Steiner | Baseline, Weeks 2, 4, 6, 8, 10, 12, and 24
  A screening questionnaire that identifies premenstrual syndrome (PMS) and premenstrual dysphoric disorder (PMDD) based on the severity and impact of symptoms.
Cognitive Flexibility Scale | Baseline, Weeks 2, 4, 6, 8, 10, 12, and 24
  A self-report questionnaire that measures an individual's ability to adapt thinking and behavior in response to changing situations and demands.
Connectedness Scale | Baseline, Weeks 2, 4, 6, 8, 10, 12, and 24
  A self-report questionnaire that assesses an individual's sense of connection to others, community, and the broader world.
SETS 2012 | Baseline, Weeks 2, 4, 6, 8, 10, 12, and 24
  A self-report questionnaire that measures patients' expectations regarding the effectiveness and outcomes of a treatment.
Treatment Guess Questionnaire | Baseline, Weeks 2, 4, 6, 8, 10, 12, and 24
  A brief measure where participants indicate which treatment condition they believe they received, used to assess blinding integrity.
Change from Baseline in Systolic Blood Pressure | Baseline, Weeks 2, 4, 6, 8, 10, 12, 24
  Systolic blood pressure measured in the seated position after 5 minutes of rest Unit of Measure: mmHg
Change from Baseline in Diastolic Blood Pressure | Baseline, Weeks 2, 4, 6, 8, 10, 12, 24
  Diastolic blood pressure measured in the seated position after 5 minutes of rest. Unit of Measure: mmHg
Change from Baseline in Heart Rate | Baseline, Weeks 2, 4, 6, 8, 10, 12, 24
  Resting heart rate by pulse/monitor. Resting heart rate by pulse/monitor
Change from Baseline in Body Temperature | Baseline, Weeks 2, 4, 6, 8, 10, 12, 24
  Oral/tympanic temperature per site SOP. Unit of Measure: °C
Change from Baseline in Salivary concentration | Baseline, Weeks 2, 4, 6, 8, 10, 12, 24
  Morning salivary collected per SOP, Unit of Measure: [ng/mL / nmol/L]
Participants with treatment-emergent clinically significant laboratory abnormalities | Baseline, Weeks 2, 4, 6, 8, 10, 12, 24
  Proportion of participants with any new or worsening clinically significant abnormality in hematology or clinical chemistry panels, per site reference ranges and PI judgment (or per predefined thresholds). Unit of Measure: % participants
Emotional Go-No-Go | On 6, 12, and 24 weeks FU.
  In this task, participants respond to certain stimuli with a motor action, while in others, they must withhold a response. Previous findings indicate impaired inhibition in patients with depression, as shown in classic response inhibition tasks using faces with negative or neutral expressions.
2 Task Switching | On 6,12, and 24 weeks FU.
  A cognitive task that measures mental flexibility and executive control by requiring participants to alternate between different tasks or rules, assessing their ability to shift attention and adapt to changing demands.
ONE-BACK | On 6,12, and 24 weeks FU.
  A working memory task in which participants view a sequence of stimuli and must indicate whether the current stimulus is the same as the one immediately preceding it, assessing attention and short-term memory.
Item & Associative recognition | On 6,12, and 24 weeks FU.
  A memory task that assesses the ability to recognize previously presented items and to recall the associations between them, measuring both item memory and relational/associative memory processes.
Qualitative interview | Baseline, 6 weeks, and 24 weeks.
  A semi-structured interview designed to capture participants' experiences, perceptions, and expectations in their own words. According to the protocol, approximately one-third of the patients will be randomly selected to participate.

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Center Beer Sheva, Beersheba, Israel